CLINICAL TRIAL: NCT00779974
Title: Electromyography Evaluation of Subscapularis Function After Total Shoulder
Brief Title: Electromyography Evaluation of Subscapularis Function After Total Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, April Armstrong, Associate Professor, Milton S. Hershey Medical Center
Other Study IDs: IRB#27370
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis
Keywords: Total Shoulder Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- s/p Total Shoulder Arthroplasty: The subject population for this study consists of adult patients with a primary diagnosis of osteoarthritis who have had a total shoulder arthroplasty preformed by the PI between September 2003 through December 2007.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — For this research study each enrolled subject will have a clinical exam, including range of motion (ROM), and strength testing. The lift off and belly compression tests will be performed. An ultrasound of the shoulder will be done to determine the integrity of the subscapularis tendon. An EMG will be done to determine functionality of the subscapularis.
  Other Names: ROM; Ultrasound; EMG; Clinic Evaluation

SUMMARY:
The primary objective is to document function of the structurally intact subscapularis after total shoulder arthroplasty by using electromyography. Structural integrity of the subscapularis will be confirmed using ultrasound.

The secondary objective is to determine the diagnostic accuracy of the belly compression and lift off tests in evaluating the integrity and function of the subscapularis when compared to the ultrasound and electromyography (EMG).

This will be accomplished by enrolling and evaluating patients with a primary diagnosis of osteoarthritis who have had a total shoulder replacement preformed by the PI from September 2003 through December 2007.

DETAILED DESCRIPTION:
The functional status of the subscapularis following total shoulder arthroplasty has not been well documented. There is evidence of loss of subscapularis function shown through physical exam in up to 2/3 of patients following total shoulder arthroplasty. [1] Multiple techniques for subscapularis repair have been demonstrated with varying degrees of post operative function, ranging from 11-66% abnormal function on physical exam. [1-3] The belly compression test and the lift off test, which are the main physical exam tests used for evaluation following surgery, are of questionable reliability as indicators of the functionality of the subscapularis. [4,5] Through comparing ultrasound evidence of an intact subscapularis to physical exam findings it has been recognized that the belly compression test has low sensitivity and specificity for subscapularis integrity. [5] Internal rotation is often limited in many postoperative total shoulder patients, which could lead to false positive results. This questions the validity of the outcomes of the studies in which the standard of testing function was through exam.

Ultrasound is a reliable exam for illustration of structural damage to the subscapularis tendon but additional testing is needed to evaluate the function of the structurally intact subscapularis. [5,6] Irreparable changes in the muscle function or nerve denervation could also result in false positive belly compression and lift off tests. The ability to accurately determine the functionality of the subscapularis following total shoulder replacement is imperative to clinic management. Although studies have shown functional abnormalities through physical exam, none have documented the functional status of the subscapularis using objective means such as EMG.

ELIGIBILITY:
Inclusion Criteria:

* age >45yrs;
* primary diagnosis of osteoarthritis of the shoulder
* total shoulder replacement performed by Dr. Armstrong between September 2003 through December 2007.

Exclusion Criteria:

* Known contraindications to ultrasound and/or EMG
* Inability to provide informed consent
* History of recent trauma to the shoulder
* Typical shoulder pain
* Other suspected shoulder pathology (i.e. tumor, infection)
* Pregnancy
* Bilateral total shoulder arthroplasty

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for this study consists of adult patients with a primary diagnosis of osteoarthritis who have had a total shoulder arthroplasty preformed by the PI between September 2003 through December 2007.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to document the function of the subscapularis after total shoulder arthroplasty | end of enrollment

SECONDARY OUTCOMES:
The sensitivity and specificity of the belly compression and lift off test will be compared to the results of the ultrasound and electromyography (EMG) | end of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: April Armstrong, MD, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Herhsey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Miller SL, Hazrati Y, Klepps S, Chiang A, Flatow EL. Loss of subscapularis function after total shoulder replacement: A seldom recognized problem. J Shoulder Elbow Surg. 2003 Jan-Feb;12(1):29-34. doi: 10.1067/mse.2003.128195. PMID 12610483
- [Background] Gerber C, Yian EH, Pfirrmann CA, Zumstein MA, Werner CM. Subscapularis muscle function and structure after total shoulder replacement with lesser tuberosity osteotomy and repair. J Bone Joint Surg Am. 2005 Aug;87(8):1739-45. doi: 10.2106/JBJS.D.02788. PMID 16085613
- [Background] Ponce BA, Ahluwalia RS, Mazzocca AD, Gobezie RG, Warner JJ, Millett PJ. Biomechanical and clinical evaluation of a novel lesser tuberosity repair technique in total shoulder arthroplasty. J Bone Joint Surg Am. 2005;87 Suppl 2:1-8. doi: 10.2106/JBJS.E.00441. No abstract available. PMID 16326718
- [Background] Tokish JM, Decker MJ, Ellis HB, Torry MR, Hawkins RJ. The belly-press test for the physical examination of the subscapularis muscle: electromyographic validation and comparison to the lift-off test. J Shoulder Elbow Surg. 2003 Sep-Oct;12(5):427-30. doi: 10.1016/s1058-2746(03)00047-8. PMID 14564261
- [Background] Armstrong A, Lashgari C, Teefey S, Menendez J, Yamaguchi K, Galatz LM. Ultrasound evaluation and clinical correlation of subscapularis repair after total shoulder arthroplasty. J Shoulder Elbow Surg. 2006 Sep-Oct;15(5):541-8. doi: 10.1016/j.jse.2005.09.013. Epub 2006 Jul 27. PMID 16979047
- [Background] Sperling JW, Potter HG, Craig EV, Flatow E, Warren RF. Magnetic resonance imaging of painful shoulder arthroplasty. J Shoulder Elbow Surg. 2002 Jul-Aug;11(4):315-21. doi: 10.1067/mse.2002.124426. PMID 12195247